CLINICAL TRIAL: NCT07255937
Title: Post Market Clinical Follow up Study to Confirm the Ongoing Safety and Performance of a Debridement Pad in Superficial, Chronic and Acute Wounds
Brief Title: PMCF Study of Debridement Pad
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Debridement Pad 001
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Ulcers; Venous Leg Ulcer; Arterial Leg Ulcer; Pressure Ulcer; Postoperative Wound Healing; Traumatic Wounds; Surgical Wounds; Burns and Scalds
MeSH Terms: conditions — Varicose Ulcer; Pressure Ulcer; Surgical Wound; Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Device: Debridement Pad

INTERVENTIONS:
Device: Debridement Pad — Study device

SUMMARY:
The design of the study is a clinical trial of Debridement Pad in subjects with superficial, chronic and acute wounds consisting of Diabetic ulcers, Arterial and Venous Leg ulcers, Pressure ulcers, Postoperative wounds healing by secondary intention, traumatic or surgical wounds and burns and scalds. The performance data from this study will support clinically meaningful rates of successful improvement in wound bed condition immediately after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 years or above.
* Patients who can understand and give informed consent to take part in the study.
* Have one or more of the following wounds: Diabetic ulcers, Arterial and Venous Leg ulcers, Pressure ulcers, Postoperative wounds healing by secondary intention, traumatic and surgical wounds, and burns and scalds
* Wounds that require debridement due to the presence of slough debris/fibrous tissue ,hyperkeratotic debris and dried exudate on the peri wound skin.
* Wounds with both serous crusts and healthy tissue.
* Minimum of 30% of the wound covered by debris, necrosis or slough.
* Wound Size > 4cm2

Exclusion Criteria:

* Patients who are known to be non-compliant with medical treatment
* Patients who are known to be sensitive to any of the device components such as polyester.
* Subject has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with their ability to participate in the study.
* Subject is currently enrolled in another clinical study, or has completed a clinical study less than 30 days prior to enrolment.
* Symptoms & signs of systemic and / or spreading wound infection (including erythema and fever).
* Severe pain (level 7 or higher on a 0-10 VAS or hyperaesthesia in the wound area).
* Subjects who in the view of the investigator might not be suitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Performance of the Debridement Pad | From baseline to immediately after treatment
  Performance of the Debridement Pad on Diabetic ulcers, Arterial and Venous Leg ulcers, Pressure ulcers, Postoperative wounds healing by secondary intention, traumatic and surgical wounds, and burns and scalds. Success will be determined by the following:
  1. Change of wound bed condition from baseline (pre debridement) to assessment immediately after the use of the debridement pad as defined as
  a. Percentage reduction of wound coverage of visible debris/necrosis/slough from the wound bed at baseline assessment and after procedure.

SECONDARY OUTCOMES:
Safety by adverse events | From baseline to immediately after treatment
  Safety will be evaluated as incidence of device-related adverse events
Time recorded for procedure | From baseline to immediately after treatment
  Time recorded for the debridement procedure
Removal of debris | From baseline to immediately after treatment
  Debris/necrosis/slough absorbed/ removed by the Debridement pad.
Pain during procedure | From baseline to immediately after treatment
  Pain during the debridement procedure time frame assessed after procedure using the Visual Analogue scale.
Overall clinician satisfaction | From baseline to immediately after treatment
  Clinician satisfaction with the device (conformability, ease of use, use of both sides, softness, integrity) will be assessed using a Likert-type scale.
Patient tolerability | From baseline to immediately after treatment
  Tolerability of the patient assessed by the clinician (assessing discomfort, pressure, burning sensation, Pain, irritation of peri wound skin, swelling and redness), assessed using a Likert-type scale.
Device use wet or dry | From baseline to immediately after treatment
  Use of the device when wet or dry (Specified, assessed using a Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Castan, PhD, Principal Investigator — Hospital Carlos III
Locations (1):
- Clínica Cres, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No